CLINICAL TRIAL: NCT06936345
Title: EVALUATION OF EFFECTIVE METHODS IN THE TREATMENT OF RESIDUAL DIZZINESS AFTER BPPV: A PARTIALLY RANDOMIZED CONTROLLED CLINICAL STUDY
Brief Title: Effective Treatments for Dizziness After BPPV: A Clinical Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Kerem Ersin, Dr., Medipol University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E-10840098-772.02-5857
Record Dates: First submitted 2025-04-13; First posted 2025-04-20 (Actual); Last update posted 2025-04-20 (Actual); Status verified 2025-04

CONDITIONS: BPPV; Residual Disease; Vestibular Disease
Keywords: Residual Dizziness; Theta Binaural Beats; Vestibular Rehabilitation; Computerized Dynamic Posturography
MeSH Terms: conditions — Neoplasm, Residual; Vestibular Diseases

STUDY DESIGN:
Intervention Model Description: Participants were assigned to one of three parallel intervention groups: Cawthorne-Cooksey Exercises (CCE), Brandt-Daroff Exercises (BDE), or CCE combined with Theta Binaural Beats (CCE+T-BB). Interventions were delivered concurrently across groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cawthorne-Cooksey Exercises (CCE) Group (Experimental): Participants in this group performed home-based Cawthorne-Cooksey vestibular rehabilitation exercises over a six-week period. Exercises were adjusted biweekly based on individual progress.
  Interventions: Behavioral: Cawthorne-Cooksey Exercises
- CCE with Theta Binaural Beats (CCE+T-BB) (Experimental): Participants followed the same six-week Cawthorne-Cooksey protocol as Arm 1, with an additional 10-minute daily Theta Binaural Beats audio session via stereo headphones.
  Interventions: Behavioral: Cawthorne-Cooksey Exercises; Other: Theta Binaural Beats
- Brandt-Daroff Exercises (BDE) Group (Active Comparator): Participants performed traditional Brandt-Daroff Exercises three times daily for four weeks. Exercises were done at home using video instructions and monitored weekly.
  Interventions: Behavioral: Brandt-Daroff Exercises

INTERVENTIONS:
Behavioral: Cawthorne-Cooksey Exercises — A set of vestibular rehabilitation exercises aimed at improving balance and reducing dizziness through repeated head and body movements, delivered via home-based digital instructions.
  Arms: CCE with Theta Binaural Beats (CCE+T-BB); Cawthorne-Cooksey Exercises (CCE) Group
Behavioral: Brandt-Daroff Exercises — A traditional home-based vestibular exercise program for treating positional dizziness, involving repetitive lateral head movements performed daily.
  Arms: Brandt-Daroff Exercises (BDE) Group
Other: Theta Binaural Beats — A digital auditory stimulation using two tones of slightly different frequencies to create a theta-frequency beat, intended to modulate anxiety and enhance vestibular rehabilitation effects.
  Arms: CCE with Theta Binaural Beats (CCE+T-BB)

SUMMARY:
This clinical study aimed to evaluate how effective vestibular rehabilitation therapy (VRT) and Theta Binaural Beats (T-BB) are in reducing dizziness and anxiety in patients who continue to feel unsteady after successful treatment for a common inner ear condition called BPPV. A total of 56 adult patients were divided into three groups, each receiving different types of home-based exercises: Cawthorne-Cooksey Exercises (CCE), Brandt-Daroff Exercises (BDE), or CCE combined with T-BB. The study measured both physical balance and emotional symptoms such as anxiety. Results showed that all treatments helped, but patients who received CCE with T-BB showed the most improvement in both balance and anxiety levels. The findings suggest that combining physical and audio-based therapy may be especially helpful for people with ongoing dizziness after BPPV.

DETAILED DESCRIPTION:
Residual dizziness (RD) is a common yet often overlooked condition that can persist after successful canalith repositioning procedures (CRP) for benign paroxysmal positional vertigo (BPPV). Despite the resolution of vertigo, many patients continue to report imbalance and anxiety, which may affect their quality of life. This study investigated whether vestibular rehabilitation therapies-specifically Cawthorne-Cooksey Exercises (CCE), Brandt-Daroff Exercises (BDE), and CCE combined with Theta Binaural Beats (CCE+T-BB)-could improve balance and reduce anxiety in patients experiencing RD.

Fifty-six adults aged 18-60 who reported dizziness for at least 20 days after CRP were enrolled. Participants were assigned to one of the three intervention groups based on auditory sensitivity. The interventions were home-based, guided by digital content through the Moodle platform, and lasted four to six weeks depending on the protocol. The CCE+T-BB group also received 10-minute daily auditory stimulation designed to modulate brainwave activity and support emotional regulation.

The study used both objective (Sensory Organization Test - SOT) and subjective (Dizziness Handicap Inventory - DHI, State-Trait Anxiety Inventory - STAI) tools to assess outcomes before and after the interventions. All groups showed improvements, but the CCE+T-BB group demonstrated superior gains in balance, especially under visually and vestibular-dependent conditions. Both CCE-based groups had significant reductions in trait and state anxiety, while the BDE group only showed improvement in trait anxiety.

These findings suggest that structured vestibular rehabilitation improves balance and reduces anxiety in patients with residual dizziness. Furthermore, adding auditory neuromodulation (T-BB) to CCE may enhance postural adaptation and emotional regulation, supporting a multimodal, non-pharmacological approach to RD management. This research represents the first clinical evaluation of Theta Binaural Beats as an adjunct to vestibular therapy and offers a promising direction for personalized rehabilitation.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with unilateral posterior canal benign paroxysmal positional vertigo (BPPV)
* Successfully treated with canalith repositioning procedures (CRP)
* Experiencing persistent dizziness or imbalance lasting at least 20 days after CRP
* Able and willing to perform home-based vestibular rehabilitation exercises
* Provided informed consent to participate in the study

Exclusion Criteria:

* Presence of other vestibular or neurological disorders (e.g., Meniere's disease, multiple sclerosis)
* History of psychiatric conditions that may interfere with participation
* Use of medications affecting vestibular function or anxiety within the last 4 weeks
* Conductive or sensorineural hearing loss
* Cognitive impairment or inability to follow digital instructions
* Previous participation in vestibular rehabilitation within the past 6 months

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2023-12-01 (Actual); Primary Completion 2025-01-01 (Actual); Study Completion 2025-01-01 (Actual)

PRIMARY OUTCOMES:
Change in Sensory Organization Test (SOT) Scores from Baseline to Post-Intervention | Baseline and Week 4/6
  The Sensory Organization Test (SOT) is a computerized dynamic posturography tool used to assess balance performance under varying sensory conditions. The Composite Score is derived from multiple stance conditions that challenge somatosensory, visual, and vestibular input. Higher scores indicate better postural stability. Scores range from 0 to 100, where a score of 100 reflects perfect stability. The primary outcome is the change in Composite Score between the baseline (pre-intervention) and post-intervention assessments.

SECONDARY OUTCOMES:
Change in Dizziness Handicap Inventory (DHI) Total and Subscale Scores from Baseline to Post-Intervention | Baseline and Week 4/6
  The Dizziness Handicap Inventory (DHI) is a 25-item questionnaire measuring the self-perceived impact of dizziness on daily life. It includes three subscales: Functional, Emotional, and Physical. Each item is scored from 0 (no handicap) to 4 (maximum handicap), and the total score ranges from 0 to 100. Higher scores indicate more severe dizziness-related disability. The outcome measure will capture changes in total and subscale scores from baseline to after the intervention.
Change in State-Trait Anxiety Inventory (STAI) Scores from Baseline to Post-Intervention | Baseline and Week 4/6
  The STAI consists of two subscales measuring state anxiety (STAI-I) and trait anxiety (STAI-II), each containing 20 items scored on a 4-point Likert scale. Total scores for each subscale range from 20 to 80, with higher scores reflecting greater anxiety. This outcome measure assesses changes in both STAI-I and STAI-II scores between baseline and post-intervention evaluations.

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul Medipol University, Istanbul, Beykoz, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data (IPD) due to privacy concerns and the absence of institutional data-sharing agreements. Additionally, the nature of the intervention and follow-up data limits the feasibility of anonymized sharing.